CLINICAL TRIAL: NCT03979651
Title: MEK and Autophagy Inhibition in Metastatic/Locally Advanced, Unresectable Neuroblastoma RAS (NRAS) Melanoma: A Phase Ib/II Trial of Trametinib Plus Hydroxychloroquine in Patients With NRAS Melanoma
Brief Title: MEK and Autophagy Inhibition in Metastatic/Locally Advanced, Unresectable Neuroblastoma RAS (NRAS) Melanoma
Acronym: CHLOROTRAMMEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL19_0115; 2019-001399-13 (EudraCT Number)
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Metastatic NRAS Melanoma
Keywords: MEK inhibitor; Autophagy inhibition; Metastatic NRAs Melanoma
MeSH Terms: interventions — trametinib; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients with NRAS Melanoma (Dose 1) (Experimental): Patients with NRAS Melanoma receiving the 1st dose of the treatment (400 milligrams)
  Interventions: Drug: Trametinib plus hydroxychloroquine in patients with NRAS Melanoma (Dose 1)
- Patients with NRAS Melanoma (Dose 2) (Experimental): Patients with NRAS Melanoma receiving the 2nd dose of the treatment (800 milligrams)
  Interventions: Drug: Trametinib plus hydroxychloroquine in patients with NRAS Melanoma (Dose 2)
- Patients with NRAS Melanoma (Dose 3) (Experimental): Patients with NRAS Melanoma receiving the 3rd dose of the treatment (600 milligrams twice a day)
  Interventions: Drug: Trametinib plus hydroxychloroquine in patients with NRAS Melanoma (Dose 3)

INTERVENTIONS:
Drug: Trametinib plus hydroxychloroquine in patients with NRAS Melanoma (Dose 1) — Standard dosing of trametinib at 2 milligrams (mg) by mouth once a day, with an escalation of hydroxychloroquine.
  The escalation of hydroxychloroquine will be decided by a 3+3 design with the goal of estimating the Maximum Tolerated Dose (MTD) of trametinib plus hydroxychloroquine. A cycle of treatment will last 28 days. Patients will be evaluated weekly during the first cycle of treatment.
  • Level -1 = Hydroxychloroquine 400 mg by mouth once a day
  Arms: Patients with NRAS Melanoma (Dose 1)
Drug: Trametinib plus hydroxychloroquine in patients with NRAS Melanoma (Dose 2) — Standard dosing of trametinib at 2 milligrams (mg) by mouth once a day, with an escalation of hydroxychloroquine.
  The escalation of hydroxychloroquine will be decided by a 3+3 design with the goal of estimating the Maximum Tolerated Dose (MTD) of trametinib plus hydroxychloroquine. A cycle of treatment will last 28 days. Patients will be evaluated weekly during the first cycle of treatment.
  • Level 1 (starting dose) = Hydroxychloroquine 800 mg by mouth once a day
  Arms: Patients with NRAS Melanoma (Dose 2)
Drug: Trametinib plus hydroxychloroquine in patients with NRAS Melanoma (Dose 3) — Standard dosing of trametinib at 2 milligrams (mg) by mouth once a day, with an escalation of hydroxychloroquine.
  The escalation of hydroxychloroquine will be decided by a 3+3 design with the goal of estimating the Maximum Tolerated Dose (MTD) of trametinib plus hydroxychloroquine. A cycle of treatment will last 28 days. Patients will be evaluated weekly during the first cycle of treatment.
  • Level 2 = Hydroxychloroquine 600 mg by mouth two times a day
  Arms: Patients with NRAS Melanoma (Dose 3)

SUMMARY:
Patients with metastatic Neuroblastoma RAS (NRAS) melanoma are currently treated with first line immune checkpoint inhibitors (nivolumab, pembrolizumab). Thus far, no targeted therapy has been approved in NRAS mutated melanoma as a second line treatment, because although the use of a MEK inhibitor (binimetinib) alone was superior to the gold standard chemotherapy (dacarbazine) in a phase 3 trial, the progression free survival gain was very modest.

In vitro and in vivo work from the study team's lab (McMAHON, Huntsman Cancer Institute (HCI), Salt Lake City), as well as, Ravi Amaravardi and Jean Mulchey-Levy suggests that the activation of autophagy is a mechanism of resistance to BRAF and MEK inhibitors in RAS and RAF mutated cancers, such as melanoma, pediatric brain tumors and pancreatic adenocarcinoma. The study team has shown in vivo, in four different NRAS mutated melanoma Patient Derived Xenograft (PDX) models that the combination of the MEK inhibitor trametinib and the autophagy inhibitor chloroquine results in a more dramatic tumor regression and inhibition than trametinib or chloroquine used as single agents (Nat Med. 2019 Apr;25(4):620-627. doi: 10.1038/s41591-019-0367-9. Epub 2019 Mar 4). In two of the PDX models, the combination resulted in almost complete tumor regression (quasi disappearance) that was not observed in the single agent treatment arms.

Trametinib (MEKINISTR) is an orally available MEK inhibitor that is currently approved in combination with the BRAF inhibitor dabrafenib (TAFINLARR) to treat BRAF mutated metastatic melanoma at the standard dosing of 2 milligrams (mg) once a day. Hydroxychloroquine (PLAQUENILR) is an orally available autophagy inhibitor that has been used for many years to treat autoimmune diseases like lupus, sarcoidosis and rheumatoid arthritis at the standard dosing of 400-600mg/day. For this study, the investigating team would like to evaluate the safety and tolerability of the combination of hydroxychloroquine and trametinib in a phase I trial in patients with NRAS mutated metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic or locally advanced unresectable malignant melanoma with an activating NRAS mutation.
2. Available archival tissue, or if not, the patient is willing to provide a baseline tumor biopsy
3. Patient must have progressed during or after a first line treatment by immunotherapy (ipilimumab, pembrolizumab, nivolumab).

   * Progression will be confirmed by two consecutive Computed Tomography (CT) assessements separated for at least 4 weeks.
   * Inclusion is possible if patients progress during an adjuvant treatment by immunotherapy or if they progress less than six months after adjuvant treatment discontinuation.
   * If patients progress six months after adjuvant treatment discontinuation, they have to be treated by a second line of immunotherapy before they can be included in the trial.
4. Patient age at least 18 years old
5. Patient Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1.
6. Patient able to provide informed consent and sign approved consent forms to participate in the study and provide tumor samples
7. Patient willing and able to comply with all study procedures and able to take oral medications.
8. Patients must be willing and able to undergo skin or tumor biopsies according to the institute's own guidelines, the study protocol and requirements for such procedures.
9. Patients must have measurable disease as defined by RECIST version 1.1 criteria
10. Adequate bone marrow, renal and liver function determined biologically:

    * Hematologic: Absolute Neutrophil Count (ANC) ≥1.5x10e9 per Liter, platelet count ≥100 x10e9 per Liter, and hemoglobin ≥9grams/deciLiter
    * Hepatic: total bilirubin level ≤1.5 times the Upper Limit of the Normal (ULN) range (except subjects with Gilbert's Syndrome who must have normal direct bilirubin) and Aspartate aminotransferase (ASAT) and Alanine Aminotransferase (ALAT) levels ≤3 ULN. For patients with metastatic disease to the liver allow levels ≤5 ULN
    * Renal: estimated creatinine clearance ≥50ml/min according to the Cockcroft-Gault formula (or local institutional standard method).
    * Albumin ≥ 27 g/l
11. Adequate cardiac function determined by a pre-treatment Electrocardiogram (EKG) and cardiac ultra-sound.

    * Corrected QT (QTc) interval ≤ 450 ms for the male population and ≤ 470ms for the female population
    * Left ventricular ejection fraction (LVEF) ≥50%
12. Women of childbearing potential must have a negative serum or urine pregnancy test at screening.
13. Both male and female patients must agree to the use of 2 methods of contraception, with one method being highly effective and the other being either highly effective or less effective throughout the study and for at least 4 months after last study treatment administration if the risk of conception exists.
14. Women of childbearing potential who are continuously not heterosexually active are exempt from contraceptive requirements. However, women of childbearing who abstain from heterosexual activity on a continuous basis must still undergo pregnancy testing as described in this protocol.

Exclusion Criteria:

1. Prior to the first dose of study treatment patient who received systemic antineoplastic therapy (including unconjugated therapeutic antibodies and toxin immunoconjugates) or any investigational therapy within 4 weeks (6 weeks for nitrosurea or mitomycin-C, antibodies like ipilimumab, pembrolizumab and nivolumab) or within 7-half lives of the investigational therapy prior to starting study treatment, whichever is longer.
2. Patient received radiotherapy within 2 weeks prior to the first dose of study treatment except localized radiation therapy for symptomatic bone metastasis
3. Patients with multiple primary malignancies may be enrolled if nonmelanoma tumor(s) are determined stable by treating investigator and do not require active treatment.
4. Patients with symptomatic brain metastases or cranial epidural disease. Asymptomatic patients with brain metastases can be included.
5. Has retinal degenerative disease (hereditary retinal degeneration or age-related macular degeneration), history of uveitis, or history of Retinal Vein Occlusion (RVO) or any eye condition that would be considered a risk factor for RVO (e.g., uncontrolled glaucoma or ocular hypertension).
6. Current evidence of uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

   * Cardio-vascular disorders: Congestive heart failure New York Heart Association (NYHA) class 3 or 4, unstable angina, uncontrolled cardiac arrhythmias, uncontrolled hypertension. Stroke, myocardial infarction or other ischemic event within 6 months before first dose.
   * History of Glucose-6-Phosphate dehydrogenase (G6PD) deficiency
   * Patients who have neuromuscular disorders that are associated with elevated Creatine Kinase (CK)
   * Impairment of gastrointestinal function or gastrointestinal disease (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection that under the judgement of the Principal Investigator (PI) may impair absorption of study drugs)
   * Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
7. Known positive serology for Human Immunodeficiency Virus (HIV), active Hepatitis B, and/or active Hepatitis C infection.
8. Patients who have undergone major surgery ≤ 3 weeks prior to starting study drug or who have not recovered from side effects of such procedure.
9. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive Human chorionic gonadotropin (hCG) laboratory test.
10. Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study
11. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 Grade≥3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) | 28 days
  DLTs will be determined weekly during the first cycle of treatment (28 days) in order to choose the optimal dose for the phase II
Percentage of patients with a partial or complete response to treatment | 56 days
  Percentage of patients with a partial or complete response to treatment according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines version 1.1 which allows the Evaluation of the Overall Response Rate (ORR) based on 3 main criteria: patients' tumor improves ("responds"), stays the same ("stabilizes"), or worsens ("progresses") during treatment. The comparison of target lesions will be based on a Computed Tomography (CT) scan performed after two cycles of treatment (56 days) to those present on the base line CT prior to treatment initiation.

SECONDARY OUTCOMES:
Change in Median progression Free survival | at the end of 2 cycles of treatment (each cycle is 28 days), at the end of the 3rd cycle of treatment and every 12 weeks thereafter up to 12 months
  Median progression Free survival will be determined in the cohort treated by the recommended phase 2 dose (RP2D). Subjects who discontinue treatment for reasons other than disease progression will have Computed Tomography (CT) scans at the end of therapy (EOT) visit (unless their previous restaging was performed within 6 weeks).
Change in Overall Survival | at the end of 2 cycles of treatment (each cycle is 28 days), at the end of the 3rd cycle of treatment and every 12 weeks thereafter up to 12 months
  Overall Survival will be determined in the cohort treated by the recommended phase 2 dose (RP2D); Subjects who discontinue treatment for reasons other than progression will have Computed Tomography (CT) scans at the end of therapy (EOT) visit (unless their previous restaging was performed within 6 weeks).
Safety of the drug combination Trametinib and Hydroxychloroquine | 1 year
  Adverse events (AEs) and Serious Adverse Events (SAEs) according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be reported
Quantification of the autophagic substrate p62 | At Day 1 (before treatment) and Day 15 (after treatment)
  p62 will be quantified by immunohistochemistry (IHC) using a skin punch biopsy of normal tissue in patients without cutaneous metastasis.
Quantification of Microtubule-associated protein Light Chain 3 (LC3) | At Day 1 (before treatment) and Day 15 (after treatment)
  LC3 will be quantified by immunohistochemistry (IHC) using a skin punch biopsy of normal tissue in patients without cutaneous metastasis.
Quantification of p-ERK | At Day 1 (before treatment) and Day 15 (after treatment)
  p-ERK will be quantified by immunohistochemistry (IHC) using a skin punch biopsy of normal tissue in patients without cutaneous metastasis.
Quantification of the autophagic substrate p62 (cutaneous metastasis) | At Day 1 (before treatment) and Day 15 (after treatment)
  p62 will be quantified by immunohistochemistry (IHC) using a skin punch biopsy of normal tissue in patients with cutaneous metastasis.
Quantification of Microtubule-associated protein Light Chain 3 (LC3) (cutaneous metastasis) | At Day 1 (before treatment) and Day 15 (after treatment)
  LC3 will be quantified by immunohistochemistry (IHC) using a skin punch biopsy of normal tissue in patients with cutaneous metastasis.
Quantification of p-ERK (cutaneous metastasis) | At Day 1 (before treatment) and Day 15 (after treatment)
  p-ERK will be quantified by immunohistochemistry (IHC) using a skin punch biopsy of normal tissue in patients with cutaneous metastasis.
Serum trametinib and hydroxychloroquine concentrations (AUC) | Day 28
  Serum trametinib and hydroxychloroquine concentrations (AUC) will be evaluated and compared to predicted published concentrations
Changes in treatment induced immune modifications in patient blood serum | At Day 1 (before treatment), at Day 15 (after treatment), at 2 months (after treatment), and at 30 days after last treatment
  The evaluation of treatment induced immune modifications in the blood serum will be based on patient peripheral blood mononuclear cell (PBMC) collection

CONTACTS AND LOCATIONS:
Overall Officials: Amélie BOESPFLUG, MD, Principal Investigator — Hospices Civils de Lyon
Locations (5):
- France (5):
  - CHU Estaing, Clermont-Ferrand, Clermont Ferrand
  - CHU Grenoble Alpes, La Tronche, La Tronche
  - AP-HP_HOPITAL Saint Louis, Paris, Paris
  - Centre Hospitalier Lyon Sud, Lyon, Pierre-Bénite
  - INSTITUT Claudius Rigaud, Toulouse, Toulouse